## THE EFFECT OF TALOCRURAL JOINT MANIPULATION ON STATIC BALANCE IN PATIENTS WITH STROKE

NCT06523010

## STATISTICAL ANALYSIS PLAN

The data were presented as either mean and Standard deviation or median, minimum, and maximum for continuous variables. Frequency and percentage were provided for categorical variables. The normal distribution of the data was evaluated with the Shapiro-Wilk test. Depending on whether the parametric assumptions were met, intergroup comparisons of the variables were conducted using the independent t-test or the Mann-Whitney U test, while intragroup comparisons of the variables were conducted using the paired samples t-test or the Wilcoxon test. The relationship between categorical variables and outcome measures was evaluated using Spearman's rank correlation. The effect of ankle mobility and the cavitation accompanying manipulation on postural stability was evaluated using regression analysis. Statistical analysis was performed using the SPSS 27 software, with the significance level set at p<.05.